CLINICAL TRIAL: NCT04795934
Title: Multicenter Single-Blind RCT of CTIF Versus LNF For Treatment of GERD in Patients Requiring Hiatal Hernia Repair Combined With Transoral Incisionless Fundoplication Versus Laparoscopic Nissen Fundoplication for Treatment of Gastroesophageal Reflux Disease in Patients Requiring Hiatal Hernia Repair
Brief Title: Multicenter Single-Blind RCT of CTIF Versus LNF For Treatment of GERD in Patients Requiring Hiatal Hernia Repair
Acronym: CTIF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: EndoGastric Solutions (Industry); University of California, Irvine (Other); Fox Valley Surgical Associates (Unknown); University of Southern California (Other); The University of Texas Health Science Center, Houston (Other); University of Texas at Austin (Other); Institute of Esophageal and Reflux Surgery (Unknown)
Responsible Party: Principal Investigator, Omar Ghanem, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 19-005226
Record Dates: First submitted 2021-02-10; First posted 2021-03-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: GERD; Hiatal Hernia
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Who Masked: Participant
Masking Description: Measures will be taken to minimize or avoid bias in the study "masking/blinding procedures." Neither treatment groups will be advised as to which procedure (TIF or LNF) they will be receiving. Randomization assignment will be recorded in the EDC and subject tracking, but will not be recorded within the EMR to reduce clinical team exposure to their randomized status for follow-up care. Research teams will not be blinded to the randomization results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic Nissen Fundoplication (LNF) (Active Comparator): Control
  Interventions: Procedure: LAPAROSCOPIC PARAESOPHAGEAL HIATAL HERNIA REPAIR COMBINED WITH TRANSORAL INCISIONLESS FUNDOPLICATION
- Combo Transoral Incisionless Fundoplication (CTIF) (Active Comparator): Treatment
  Interventions: Procedure: LAPAROSCOPIC PARAESOPHAGEAL HIATAL HERNIA REPAIR COMBINED WITH TRANSORAL INCISIONLESS FUNDOPLICATION

INTERVENTIONS:
Procedure: LAPAROSCOPIC PARAESOPHAGEAL HIATAL HERNIA REPAIR COMBINED WITH TRANSORAL INCISIONLESS FUNDOPLICATION — LAPAROSCOPIC PARAESOPHAGEAL HIATAL HERNIA REPAIR COMBINED WITH TRANSORAL INCISIONLESS FUNDOPLICATION VERSUS LAPAROSCOPIC NISSEN FUNDOPLICATION
  Other Names: LAPAROSCOPIC NISSEN FUNDOPLICATION

SUMMARY:
This single-blind randomized control study will follow 142 subjects across 7 sites randomized on a 1:1 ratio to compare treatment efficacy and safety between TIF and LNF in GERD patients with hiatal hernia undergoing hernia repair.

ELIGIBILITY:
Inclusion Criteria:

1. 22-80 years of age
2. Subjects have GERD with hiatal hernia < 5 cm (defined as maximum ,axial height from end of the esophagus to diaphragm by any study including upper endoscopy esophagram and or at time of surgery) and Hill grade III or IV
3. Pathologic reflux while off PPI based on Lyon criteria by either of the following:

   3.1. Conclusive evidence for pathologic reflux defined as acid exposure time (AET) > 6% (worst day) or LA grade C or D esophagitis.

   3.2. Borderline evidence of pathologic reflux defined as presence of one of the following parameters: AET 4-6%, LA grade A or B.
4. Commitment to long-term study
5. Ability to give consent individually or by a legally authorized representative

Exclusion Criteria:

1. Hiatal hernia > 5 cm (defined as maximum axial height from end of the esophagus to diaphragm by any study including upper endoscopy esophagram and or at time of surgery)
2. Evidence of clinically significant major esophageal motility disorder as determined by the site primary investigator
3. Pregnancy (in females) at time of procedure
4. Previous anti-reflux procedure
5. Subjects requiring mesh treatment at time of procedure
6. At the discretion of the site PI for subject safety
7. BMI > 35 at time of surgery.
8. Prior gastric surgery that may affect ability to perform either procedure or affect normal gastric function (e.g. gastrectomy, gastric bypass, sleeve gastrectomy, pyloroplasty.
9. Severe gastroparesis

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Mean difference in HRQL score ≤ 15% | 6 months
  Hypothesis: TIF is non-inferior to LNF as measured by quality of life at 6 months post-procedure using the Gastroesophageal Reflux Disease-Health-Related Quality of Life (GERD-HRQL) score.
  GERD-HRQL Scoring Total Score: Calculated by summing the individual scores to questions 1-15.
  * Greatest possible score (worst symptoms) = 75
  * Lowest possible score (no symptoms) = 0
  Heartburn Score: Calculated by summing the individual scores to questions 1-6 .
  * Worst heartburn symptoms = 30
  * No heartburn symptoms = 0
  * Scores of ≤ 12 with each individual question not exceeding 2 indicate heartburn elimination.
  Regurgitation Score: Calculated by summing the individual scores to questions 10-15.
  * Worst regurgitation symptoms = 30
  * No regurgitation symptoms = 0
  * Scores of ≤ 12 with each individual question not exceeding 2 indicate regurgitation elimination.

SECONDARY OUTCOMES:
Change in AET | [Time Frame: 6 months]
  Upper Endoscopy with 72 Hrs BravoPH Case Report Form
Incidence of bloating | [Time Frame: 6 months]
  Dysphagia, Bloating, & Reflux Symptoms Questionnaire (DBR) Case Report Form
Incidence of dysphagia | [Time Frame: 6 months]
  Dysphagia, Bloating, & Reflux Symptoms Questionnaire (DBR) Case Report Form
Change in distensibility index of GE junction | [Time Frame: 6 months]
  Endoflip (optional) Case Report Form
Cessation of Proton Pump Inhibitor (PPI) use | [Time Frame: 6 months]
  PPI Use Questionnaire Case Report Form
Healing of esophagitis | [Time Frame: 6 months]
  Upper Endoscopy with 72 Hrs BravoPH Case Report Form assessing LA Grade system: A, B, C, or D (if present)
  Grade A One (or more) mucosal break no longer than 5 mm that does not extend between the tops of two mucosal folds Grade B One (or more) mucosal break more than 5 mm long that does not extend between the tops of two mucosal folds Grade C One (or more) mucosal break that is continuous between the tops of two or more mucosal folds but which involve less than 75% of the circumference Grade D One (or more) mucosal break which involves at least 75% of the esophageal circumference
Recurrence of hiatal hernia | [Time Frame: 6 months]
  Upper Endoscopy with 72 Hrs BravoPH Case Report Form
Hill grade of GE junction | [Time Frame: 6 months]
  Upper Endoscopy with 72 Hrs BravoPH Case Report Form
Adverse events rate | [Time Frame: 6 months]
  Adverse Event Case Report Form

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California Irvine, Irvine, California
  - University of Southern California, Los Angeles, California
  - Institute of Esophageal and Reflux Surgery, Englewood, Colorado
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - The University of Texas at Austin, Austin, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Fox Valley Surgical, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Health information may be collected from: Past, present and future medical records. Research procedures, including research office visits, tests, interviews and questionnaires. Health information will be used and/or given to others to: Do the research. Report the results. See if the research was conducted following the approved study plan, and applicable rules and regulations. Health information may be used and shared with: Mayo Clinic research staff involved in this study or clinical care. Researchers involved in this study at other institutions. The sponsor of this study and the people or groups hired by the sponsor to help perform this research. The Mayo Clinic Institutional Review Board that oversees the research. Federal and State agencies (such as the Food and Drug Administration, the Department of Health and Human Services, the National Institutes of Health and other United States agencies) or government agencies in other countries that oversee or review research.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials